CLINICAL TRIAL: NCT00393289
Title: Calcium Absorption and Retention From Marine Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KF-01270319; M182
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Calcium Metabolism
Keywords: Calcium absorption; D-vitamin status; Whole body calcium retention; Calcium intake; PTH status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Calcium controlled diet

SUMMARY:
The purpose of the study is to determine the uptake of calcium from fish bone meal from salmon and cod in 12 healthy volunteers. A test meal labelled with trace amounts of a radioactive calcium isotope (Ca47) will be given after an overnight fast and whole body retention of calcium will be measured on day 13, 21, and 24 after the test meal day.

DETAILED DESCRIPTION:
Background:

Up till now little attention has been given the exploitation of marine by-products from the fishing industry. Calcium in fish is found mainly in bone and skin. By-products from these sources are limited to production of gelatine. Small fish, which can be eaten whole with bones included, are traditionally considered to be a good source of calcium. Until recently, bioavailability of this calcium was not known. Two recent studies from Denmark have shown that the absorption of calcium from small soft-boned fish was comparable to that of skimmed milk both in rats and in humans.

Calcium fortified foods are likely to play an important role in helping consumers to achieve calcium requirements aimed at reducing the risk of developing osteoporosis. Experimental evidence show a positive effect of calcium supplementation on bone mineral accretion in children, and combined calcium and vitamin D supplementation has resulted in reduced bone loss and fracture incidence in older men and women.

This protocol describes a project on the nutritional utilisation of calcium from fish bone waste. The main objective is to maximise the use and the added value of marine by-products with special emphasis on utilisation of fish bone as a calcium source and determine its bioavailabiliy in humans.

Study design :

This study will follow a 3x7 weeks ransomised crossover design, where the calcium absorption and retention will be measured form meals labelled with 47Ca. The test meals will be digested in the morning after a 12h fast and bloodsampling. Whole body retention will be measured on day 15, 22 and 26, and calibrated against a background measurement from the day prior to ingestion of the test meal. The subjects will receive an ordinary standardised diet for 2 days prior and 3 days after the test meals. This diet will be standardised to match the subjects' individual calcium intake.

Test meals:

Two types of fish bone meal (from salmon and cod fish) and a control (CaCO3) will be tested. Amounts equivalent of 800 mg Ca will be baked into bread, which will be labelled with 47Ca and served with 500 mL of ultra pure water at the department.

Isotopes and labelling procedure:

Isotopes (47Ca) will be ordered from Risø National Laboratory, Radiation Research Department, Denmark. The department of Human Nutrition will recieve the prepared doses of isotopes the day before the test meal. A dose of 0.2 MBq/ml will be used. The doses will be used to extrinsically label the test meals by drop-wise adding 1 ml of isotope solution in the afternoon on the day before intake of test meals and stored at 5 degree C until ingested.

Since each subject will recieve labelled meals on three occasions, a total dose of 0.6 MBq will be ingested during the study.

Measurement of calcium retention:

The whole body retention of calcium will be measured with a whole body counter at the Copenhagen University Hospital, Denmark. All measurements of calcium retention will be corrected for physical decay back to the time of administration.

Chemical analyses:

Serun calcium, phosphorus and vitamin D concentrations will be determined in before each test meal. Plasma levels of PTH will be determined before the first test meal only.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* BMI: 18-18 kg/m2
* age: 18-40 years

Exclusion Criteria:

* elite athletes
* on medication
* gastrointestinal disorders, chronic diseaes
* smoking
* prior participation in radioisotpe studies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-11; Primary Completion 2006-04 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Whole body retention of calcium

SECONDARY OUTCOMES:
D-vitamin and PTH status, serum calcium and phosporus, and calcium intake

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bügel, MSc, PhD, Principal Investigator — Institute of Human Nutrition, THe Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Institute of Human Nutirtion, The Royal Veterinary and Agricultural University, Denmark, Frederiksberg, Frederiksberg C, Denmark

IPD SHARING:
Plan to Share IPD: Yes